CLINICAL TRIAL: NCT03003481
Title: Follow-up Registry to Monitor the Efficacy and Safety of the Occlutech PLD Device
Status: Completed | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2016_01
Record Dates: First submitted 2016-10-24; First posted 2016-12-28 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Mitral Paravalvular Leaks (PVL); Aortic Paravalvular Leaks (PVL)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Collect patient data and to monitor the clinical use (safety and efficacy) of the device

ELIGIBILITY:
Inclusion criteria:

- Patients with PVL associated hemolysis, recurrent blood transfusions, or hemodynamically significant heart failure

Exclusion criteria

The device is contraindicated for patients known to have any of the following:

* Known coagulation dysfunction
* Leak reversal with separate or significant residual or recurrent leak
* Acute infection
* Known intra-cardiac thrombi
* Recent pelvic venous thrombosis
* Recent myocardial infarction or a surgical bypass operation in the last 30 days
* If adequate oral anticoagulation therapy / antiplatelet aggregation inhibition is not possible post-procedurally
* Intolerance of contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic or mitral PVL
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2016-10; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Proper closure of the PVL (defined as Reduction in paravalvular regurgitation of ≥ one grade as assessed by echocardiography pre vs post implantation) and/or reduction in the number of hemolysis related transfusions. | 6 month following implantation
Absence of device -and/or procedure-related Serious Adverse Events (SAEs) including deaths, stroke (ischemic stroke that occurs within 24 hours following implantation), systemic embolism or device embolizations. | 6 month following implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Bergamo, Italy